CLINICAL TRIAL: NCT01210859
Title: Effects of Antimuscarinic Drugs on OAB Symptoms After Insertion of Ureteral Stents
Brief Title: Effects of Antimuscarinic Drugs on Overactive Bladder (OAB) Symptoms After Insertion of Ureteral Stents
Status: Withdrawn | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: URSTDETRUSITOL
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Overactive Bladder
Keywords: detrusitol; overactive; bladder; ureteral; stents
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ureteral stents Detrusitol treatment Lyfestyle outcome: Ureteral stents Detrusitol treatment Lyfestyle outcome

SUMMARY:
The purpose of this study is to check whether antimuscarinics that usually broadly used in the treatment of overactive bladder symptoms are effective in the treatment of those symptoms after insertion of ureteral stents. In order to study the efficacy of the treatment of OAB symptoms in stented patients the investigator will use a suitable questionnary.

ELIGIBILITY:
Inclusion Criteria:

* everyone who underwent ureteral stent insertion and started the treatment with detrusitol

Exclusion Criteria:

* adverse affects of detrusitol or unwillness of the patient to continue the treatment with detrusitol, cronic renal or hepatic failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients which underwent ureteral stent insertion
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)